CLINICAL TRIAL: NCT00632424
Title: A Phase 1 Study of Ixabepilone Administered as 3 Oral Doses Each Separated by 6 Hours Every 21 Days in Subjects With Advanced Cancer
Brief Title: Phase 1 Trial of Oral Ixabepilone
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business Objectives Changed
Sponsor: R-Pharm (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-149
Record Dates: First submitted 2008-03-03; First posted 2008-03-10 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — ixabepilone; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Ixabepilone (oral formulation)

INTERVENTIONS:
Drug: Ixabepilone (oral formulation) — Capsules, Oral, Dose escalating (Phase 1), 3 doses on 1 day every 3 weeks, until disease progression or unacceptable toxicity
  Other Names: IXEMPRA; BMS-247550

SUMMARY:
This Phase 1 study of oral ixabepilone given every 6 hours for 3 doses on Day 1, every 21 days, was a dose-finding study designed to determine the maximum tolerated dose (MTD) and safety of this dosing schedule in participants with advanced cancer

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 or older
* Histologically or cytologically confirmed diagnosis of solid tumor malignancy
* Measurable or non-measurable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) criteria
* Karnofsky Performance Status (KPS) of 70-100
* Recovered from toxicities resulting from previous therapies

Exclusion Criteria:

* More than 3 prior cytotoxic regimens in the metastatic setting
* Current or recent gastrointestinal (GI) disease that would impact the absorption of study drug
* Inability to swallow whole capsules
* Inadequate hepatic and renal function
* Function exposure to any epothilone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Stanford University, Stanford, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 participants enrolled in this study; five participants were never treated due to not meeting study criteria (n=4) and withdrawal of consent (n=1).
Groups:
- All Treated Participants: Ixabepilone was given as 3 oral doses separated by 6 hours at 30 mg, 40 mg, or 50 mg doses every 6 hours for 3 total doses on Day 1 of a 21-day cycle.
Period: Overall Study
Arm/Group | All Treated Participants
Started | 18
Completed | 0
Not Completed | 18
Not completed — Disease Progression | 17
Not completed — Study Drug Toxicity | 1

BASELINE CHARACTERISTICS:
Groups:
- Ixabepilone 90 mg/Day: The starting dose level was 30 mg/dose for ixabepilone given as 3 oral doses separated by 6 hours (30 mg every 6 hours for 3 doses) on Day 1 of a 21-day cycle for a total dose of 90 mg per cycle.
- Ixabepilone 120 mg/Day: Participants received 40 mg/dose for ixabepilone given as 3 oral doses separated by 6 hours (40 mg every 6 hours for 3 doses) on Day 1 of a 21-day cycle for a total dose of 120 mg per cycle.
- Ixabepilone 150 mg/Day: Participants received 50 mg/dose for ixabepilone given as 3 oral doses separated by 6 hours (50 mg every 6 hours for 3 doses) on Day 1 of a 21-day cycle for a total dose of 150 mg per cycle.
- Total: Total of all reporting groups
Arm/Group | Ixabepilone 90 mg/Day | Ixabepilone 120 mg/Day | Ixabepilone 150 mg/Day | Total
Number analyzed (Participants) | 3 | 9 | 6 | 18
Age, Continuous [Median (Full Range); unit: years] | 59.0 [47.0 to 70.0] | 69.0 [39.0 to 75.0] | 56.0 [27.0 to 60.0] | 59.0 [27.0 to 75.0]
Age, Customized [Number; unit: participants]
  Greater than, equal to 65 years | 1 | 5 | 0 | 6
  Less than 65 years | 2 | 4 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 3 | 10
  Male | 1 | 4 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Dose-Limiting Toxicity (DLT)
Description: DLT: any of the following, considered related to ixabepilone, occurring in Cycle 1: Absolute neutrophil count (ANC) <500 cells/mm^3 for ≥5 consecutive days or febrile neutropenia of any duration; Grade(Gr)4 thrombocytopenia <25,000 cells/mm^3 or Gr3 with bleeding requiring platelet transfusion; Gr3/4 nausea, vomiting, or diarrhea despite use of adequate intervention, fatigue, any other clinically significant drug-related ≥Gr 3 non-hematologic toxicity, delayed recovery (to Gr ≤1 or baseline, except alopecia) from toxicity which delays initiation of Cycle 2 by ≥3 weeks.
Time Frame: During Cycle 1 (Day 0 through Day 21)
Population: All participants who received at least one dose of ixabepilone.
Measure: Number; unit: participants
Arm/Group | Ixabepilone 90 mg/Day | Ixabepilone 120 mg/Day | Ixabepilone 150 mg/Day
Number analyzed (Participants) | 3 | 9 | 6
participants
  ANC <500 cells/mm^3 for ≥5 consecutive days | 0 | 0 | 0
  Grade 4 febrile neutropenia | 0 | 1 | 0
  Grade 4 neutropenic sepsis | 0 | 0 | 1
  Grade 4 thrombocytopenia <25000 cells/mm^3 | 0 | 0 | 0
  Grade 3 thrombocytopenia with bleeding episode | 0 | 0 | 0
  Grade 3/4 nausea | 0 | 0 | 0
  Grade 3/4 vomiting | 0 | 0 | 0
  Grade 3/4 diarrhea | 0 | 0 | 0
  Fatigue | 0 | 0 | 0
  Drug-related ≥3 non-hematologic toxicity | 0 | 0 | 0
  Delayed recovery from drug-related toxicity | 0 | 0 | 0

2. Primary Outcome: Ixabepilone Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (R2PD)
Description: The MTD was defined as the maximum dose which could be given to 6 participants such that not more than 1 participant experienced a DLT (or fewer than one-third if there were more than 6 treated participants) with at least 2 participants experiencing a DLT at the next higher dose level. The R2PD was to be based on the MTD and the assessment of any relevant chronic toxicities.
Time Frame: At the end of Cycle 1 (21 days).
Population: Due to early study discontinuation, the MTD and RP2D of oral ixabepilone at the scheduled doses used in this study were not determined
Arm/Group | All Treated Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Event (AE), AE Leading to Discontinuation, Treatment-related AE, Treatment-related AE Leading to Discontinuation (DC), Most Common Treatment-Related Nonhematologic AE (>25%), Serious AE (SAE), or Treatment-related SAE
Description: AEs graded according to Common Terminology Criteria Version 3.0 (CTC v 3.0). AE=any new untoward medical occurrence or worsening of a pre-existing medical condition not necessarily having a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization/causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, or is an important medical event.
Time Frame: From first study drug administration through 30 days post dose
Population: All participants who received at least one dose of ixabepilone.
Measure: Number; unit: participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 18
participants
  Grade (Gr) 1 (mild) AE | 2
  Gr 2 (moderate) AE | 7
  Gr 3 (severe) AE | 5
  Gr 4 (life-threatening, [LT]) AE | 2
  Gr 5 (death) AE | 1
  All AEs | 17
  Gr 4 (LT) AE Leading to Discontinuation (DC) | 1
  All AEs Leading to DC | 1
  Gr 1 (mild) Treatment-related AE | 7
  Gr 2 (moderate) Treatment-related AE | 5
  Gr 3 (severe) Treatment-related AE | 2
  Gr 4 (LT) Treatment-related AE | 2
  All Treatment-related AEs | 16
  Gr 3 (severe) SAE | 2
  Gr 4 (LT) SAE | 2
  Gr 5 (death) SAE | 1
  All SAEs | 5
  Gr 4 (LT) Treatment-related SAE | 2
  All Treatment-related SAE | 2

4. Secondary Outcome: Number of Participants With Most Common Treatment-Related Nonhematologic AEs (>25%)
Description: as for outcome 3
Time Frame: From first study drug administration through 30 days post dose
Population: All participants who received at least one dose of ixabepilone.
Measure: Number; unit: participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 18
participants
  Gr 1 (mild) Fatigue | 4
  Gr 2 (moderate) Fatigue | 3
  Gr 4 (LT) Fatigue | 1
  All Fatigue | 8
  Gr 1 (mild) Nausea | 7
  All Nausea | 7

5. Secondary Outcome: Number of Participants With Hematology Laboratory Abnormalities
Description: Laboratory results were graded according to CTC v 3.0. Hematology laboratory evaluations included absolute neutrophil count (ANC), white blood cell count (WBC), platelets (PLT), and hemoglobin (HGB).
Time Frame: From first study drug administration through 30 days post dose
Population: All participants who received at least one dose of ixabepilone.
Measure: Number; unit: participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 18
participants
  Gr 0 (no abnormality) WBC | 4
  Gr 1 (mild) WBC | 5
  Gr 2 (moderate) WBC | 5
  Gr 3 (severe) WBC | 1
  Gr 4 (LT) WBC | 3
  Gr 0 (no abnormality) ANC | 8
  Gr 1 ANC | 3
  Gr 2 (moderate) ANC | 2
  Gr 3 (severe) ANC | 3
  Gr 4 (LT) ANC | 2
  Gr 0 (no abnormality) PLT | 14
  Gr 1 (mild) PLT | 3
  Gr 4 (LT) PLT | 1
  Gr 1 (mild) HGB | 10
  Gr 2 (moderate) HGB | 8

6. Secondary Outcome: Number Of Participants With Liver Function and Renal Laboratory Abnormalities
Description: Laboratory results were graded according to CTC v 3.0. Clinical laboratory evaluations included liver function (alanine aminotransferase [ALT], Aspartate aminotransferase [AST], alkaline phosphatase, and total bilirubin), and renal function (creatinine).
Time Frame: From first study drug administration through 30 days post dose
Population: Since study NCT00632424 (CA163-149) was discontinued early due to variability in oral ixabepilone concentrations with the potential to negatively impact both safety and efficacy, liver and renal laboratory data were collected but not summarized.
Arm/Group | All Treated Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Maximum QTc Interval on Day 1 and Maximum Change From Baseline for QTc Interval
Description: QTc interval was defined as the measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle, corrected for heart rate
Time Frame: Baseline (Day -1) and Day 1
Population: Since study NCT00632424 (CA163-149) was discontinued early due to variability in oral ixabepilone concentrations with the potential to negatively impact both safety and efficacy, QTc data were collected but not analyzed.
Groups:
- Ixabepilone 30 mg/Dose: The starting dose level was 30 mg/dose for ixabepilone given as 3 oral doses separated by 6 hours (30 mg every 6 hours for 3 doses) on Day 1 of a 21-day cycle for a total dose of 90 mg per cycle.
- Ixabepilone 40 mg/Dose: Participants received 40 mg/dose for ixabepilone given as 3 oral doses separated by 6 hours (40 mg every 6 hours for 3 doses) on Day 1 of a 21-day cycle for a total dose of 120 mg per cycle.
- Ixabepilone 50 mg/Dose: Participants received 50 mg/dose for ixabepilone given as 3 oral doses separated by 6 hours (50 mg every 6 hours for 3 doses) on Day 1 of a 21-day cycle for a total dose of 150 mg per cycle.
Arm/Group | Ixabepilone 30 mg/Dose | Ixabepilone 40 mg/Dose | Ixabepilone 50 mg/Dose
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: PK: Mean Plasma Concentration Of Ixabepilone By Nominal Collection Time
Description: Pharmacokinetics (PK) of ixabepilone were derived from plasma concentration versus time data. Individual patient PK parameter values were derived by standard non-compartmental methods by a validated pharmacokinetic analysis program. PK parameters include Cmax (maximum plasma concentration), Cmin (minimum plasma concentration), Tmax (time of maximum plasma concentration), AUC (0-TAU) (area under the curve in one dosing interval), T-half (plasma half-life).
Time Frame: Time 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 12.5, 13, 14, 15, 16, 17, 18, 20, 48, 72, and 168 hours post dose
Population: Number of Participants Analyzed =All participants who received any treatment with ixabepilone and had adequate concentration profiles, n=all participants who received ixabepilone and had adequate concentration profiles at the specified time point. Cmax, Cmin, Tmax, AUC (0-TAU), and T-half were not calculated.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Ixabepilone 120 mg/Day: Participants received 40 mg/dose for ixabepilone given as 3 oral doses separated by 6 hours (40 mg every 6 hours for 3 doses on Day 1 of a 21-day cycle for a total dose of 120 mg per cycle.
- Ixabepilone 150 mg/Day: Participants received 50 mg/dose for ixabepilone given as 3 oral doses separated by 6 hours (50 mg every 6 hours for 3 doses on Day 1 of a 21-day cycle for a total dose of 150 mg per cycle.
Arm/Group | Ixabepilone 90 mg/Day | Ixabepilone 120 mg/Day | Ixabepilone 150 mg/Day
Number analyzed (Participants) | 3 | 9 | 6
ng/ml
  Time 0 hours (hrs) | 0 (0) | 0 (0) | 0 (0)
  Time 0.5 hrs (n=1, n=1, n=1) | 2.77 (0) | 11.46 (0) | 7.86 (0)
  Time 1 hrs (n=1, n=5, n=4) | 9.31 (0) | 19.93 (21.3) | 41.82 (52.44)
  Time 2 hrs (n=2, n=6, n=n=6) | 29.67 (29.49) | 73.57 (81.25) | 104.91 (52.99)
  Time 3 hrs (n=3, n=8, n=6) | 52.75 (54.89) | 56.2 (33.30) | 124.51 (66.16)
  Time 4 hrs (n=3, n=8, , n=6) | 24.18 (13.62) | 30.23 (21.80) | 52.16 (31.23)
  Time 5 hrs (n=3, n=8, n=6) | 16.64 (9.66) | 22.24 (18.62) | 36.54 (21.13)
  Time 6 hrs (n=3, n=8, n=6) | 12.84 (7.81) | 17.75 (15.92) | 32.08 (20.15)
  Time 8 hrs (n=3, n=8, n=6) | 11.19 (3.87) | 32.50 (33.33) | 104.54 (122.82)
  Time 12 hrs (n=3, n=9, n=6) | 26.76 (35.20) | 24.84 (38.33) | 49.41 (26.57)
  Time 12.5 hrs (n=3, n=9, n=6) | 24.24 (30.31) | 22.58 (35.24) | 78.35 (102.94)
  Time 13 hrs (n=3, n=9, n=6) | 17.63 (20.47) | 25.94 (30.20) | 103.24 (166.47)
  Time 14 hrs (n=3, n=9, n=6) | 19.6 (24.98) | 52.17 (51.73) | 59.02 (74.01)
  Time 15 hrs (n=3, n=9, n=6) | 18.52 (23.07) | 39.52 (29.80) | 86.30 (134.08)
  Time 16 hrs (n=3, n=9, n=6) | 27.37 (23.34) | 43.62 (37.63) | 93.53 (144.91)
  Time 17 hrs (n=3, n=9, n=6) | 76.63 (79.12) | 37.31 (33.27) | 116.04 (196.12)
  Time 18 hrs (n=3, n=9, n=6) | 38.32 (27.42) | 41.13 (45.41) | 94.27 (142.91)
  Time 20 hrs (n=3, n=9, n=6) | 24.71 (17.20) | 43.04 (38.39) | 89.71 (78.41)
  Time 48 hrs (n=2, n=9, n=4) | 11.77 (4.16) | 13.60 (17.77) | 24.41 (15.33)
  Time 72 hrs (n=2, n=8, n=4) | 7.20 (2.05) | 10.49 (12.68) | 14.81 (9.62)
  Time 168 hrs (n=1, n=4, n=n=4) | 3.12 (0.00) | 7.80 (7.84) | 6.28 (5.90)

9. Secondary Outcome: Best Overall Response
Description: Tumor assessment was performed according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR) = disappearance of all clinical and radiological evidence of target lesions; Partial Response (PR) = at least 30% reduction in the sum of the longest diameter of all target lesions; Progressive disease (PD) = at least 20% increase in the sum of the longest diameter of all target lesions; Stable Disease (SD) = neither PR nor PD criteria were met.
Time Frame: Tumor assessments performed on Day 1 of every other cycle of therapy, until disease progression or toxicity
Population: All treated participants who received at least one dose of ixabepilone were evaluable for tumor response.
Measure: Number; unit: participants
Arm/Group | Ixabepilone 30 mg/Dose | Ixabepilone 40 mg/Dose | Ixabepilone 50 mg/Dose
Number analyzed (Participants) | 3 | 9 | 6
participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 1 | 2 | 2
  Progressive Disease | 2 | 7 | 3
  Unable To Be Determined | 0 | 0 | 1

ADVERSE EVENTS:
Arm/Group | Ixa 90 mg/Day | Ixa 120 mg/Day | Ixa 150 mg/Day
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/9 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 8/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixa 90 mg/Day (N=3) | Ixa 120 mg/Day (N=9) | Ixa 150 mg/Day (N=6)
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 1 | 0
NEUTROPENIC SEPSIS (Infections and infestations) | 0 | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 1
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 1
CHEST PAIN (General disorders) | 1 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 1 | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixa 90 mg/Day (N=3) | Ixa 120 mg/Day (N=9) | Ixa 150 mg/Day (N=6)
DIPLOPIA (Eye disorders) | 0 | 1 | 0
EYE PAIN (Eye disorders) | 1 | 0 | 0
EYELID OEDEMA (Eye disorders) | 1 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 1 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 0 | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 1 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 0
VENA CAVA THROMBOSIS (Vascular disorders) | 0 | 0 | 1
INSOMNIA (Psychiatric disorders) | 0 | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1 | 1
TREMOR (Nervous system disorders) | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 0
DIZZINESS (Nervous system disorders) | 1 | 1 | 0
DYSGEUSIA (Nervous system disorders) | 1 | 2 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 1 | 5 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 2 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 1 | 1
DRY MOUTH (Gastrointestinal disorders) | 1 | 0 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 1 | 2
PROCTALGIA (Gastrointestinal disorders) | 0 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 1 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 3 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 1 | 0
FOLLICULITIS (Infections and infestations) | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 0 | 1 | 0
FUNGAL INFECTION (Infections and infestations) | 0 | 0 | 1
ESCHERICHIA INFECTION (Infections and infestations) | 0 | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
RENAL PAIN (Renal and urinary disorders) | 1 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 1 | 0
ANOREXIA (Metabolism and nutrition disorders) | 2 | 2 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 0 | 3 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 2 | 1
DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
SCROTAL PAIN (Reproductive system and breast disorders) | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
SINUS DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
FATIGUE (General disorders) | 3 | 4 | 4
PYREXIA (General disorders) | 0 | 1 | 0
CHEST PAIN (General disorders) | 1 | 0 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 2 | 0
TEMPERATURE INTOLERANCE (General disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The MTD of oral ixabepilone at the scheduled doses used in this study was not determined due to early study discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.